CLINICAL TRIAL: NCT00525343
Title: Avonex® Fifteen Year Long Term Follow Up of Patients With Relapsing Multiple Sclerosis: ASSessment of Drug Utilization, EaRly TreAtmeNt, and Clinical OutcomEs
Brief Title: Avonex 15 Year Long Term Follow-up Study
Acronym: 15yASSURANCE
Status: Completed | Type: Observational
Sponsor: Biogen (Industry)
Responsible Party: Pamula Foulds, Biogen Idec
Other Study IDs: 007-06-AVX
Record Dates: First submitted 2007-09-04; First posted 2007-09-05 (Estimated); Last update posted 2010-03-08 (Estimated); Status verified 2010-03

CONDITIONS: Multiple Sclerosis
Keywords: Avonex pivotal trial; Avonex; Avonex long term follow-up; Avonex outcomes
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The Avonex Fifteen-year Long-term Follow-up of Patients with Relapsing Multiple Sclerosis: ASSessment of Drug Utilization, EaRly TreAtmeNt, and Clinical OutcomEs (ASSURANCE), was a single-time-point evaluation of patients conducted 15 years after the pivotal MSCRG study, evaluated the impact of IM IFNβ-1a treatment on long-term disability and Quality of Life outcomes in patients who completed 2 years in a previous Multiple Sclerosis Collaborative Research Group (MSCRG) study.

DETAILED DESCRIPTION:
The primary objective of this study is to determine the impact of early versus delayed initiation of treatment on the long-term physical status of patients with relapsing forms of MS measured by the self-reported EDSS.

Primary endpoints for this study were as follows:

1. Changes in EDSS score from baseline for original Avonex® pivotal trial
2. Percentage of patients with EDSS scores less than or equal to 4
3. Percentage of patients with EDSS scores less than or equal to 6
4. Percentage of patients with EDSS scores less than or equal to 7

Secondary endpoints were:

1. Percentage of patients alive
2. Percentage of patients living independently
3. SF 36 Quality of Life status
4. Self-reported VAS of independence with self-care

ELIGIBILITY:
Inclusion Criteria:

1. Patients having completed at least 2 years of treatment (Avonex® or placebo) in the original Avonex® pivotal trial.
2. Subjects (or their caregivers) must be willing to complete a multi-page questionnaire.
3. Signed written informed consent form

Exclusion Criteria:

1. Unwillingness or inability to comply with the requirements of this protocol.
2. Any other reasons that, in the opinion of the Investigator, the subject is determined to be unsuitable for enrollment into this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients having completed at least 2 years of treatment (Avonex® or placebo) in the original Avonex® pivotal trial.
Sampling Method: Non-Probability Sample
Enrollment: 122 (Actual)
Dates: Start 2007-03; Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
To determine the impact of early versus delayed initiation of treatment on the long-term disability status of patients with relapsing forms of multiple sclerosis (MS) measured by the self-reported EDSS. | 15 years

SECONDARY OUTCOMES:
To determine the impact of early versus delayed initiation of treatment on patients' mortality, living independence, and quality of life. | 15 years

CONTACTS AND LOCATIONS:
Overall Officials: Pamela Foulds, MD, Study Director — Biogen
Locations (4):
- United States (4):
  - Georgetown University Medical Center, Washington D.C., District of Columbia
  - Jocab's Neurological Institute, Buffalo, New York
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Oregon Health and Science University, Portland, Oregon